CLINICAL TRIAL: NCT05042323
Title: The Landslide Disaster in Gjerdrum Municipality: Early Intervention and Health Trajectories After Mass Trauma
Brief Title: Short-term Intervention and Health Trajectories After Mass Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gjerdrum
Record Dates: First submitted 2021-03-14; First posted 2021-09-13 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2021-09

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TF-CBT-Skills (Experimental): Step 1: 4-5 sessions with stabilization/skill building Step 2: 4-5 sessions with narrative and cognitive processing
  Interventions: Behavioral: TF-CBT-Short
- TF-CBT-Narr (Active Comparator): Step 1: 4-5 sessions with narrative and cognitive processing Step 2: 4-5 sessions with stabilization/skill building
  Interventions: Behavioral: TF-CBT-Short

INTERVENTIONS:
Behavioral: TF-CBT-Short — Participants receive either 4-5 sessions of TF-CBT-Skills or TF-CBT-Narr. If the participant still has significant PTSS they are provided with step two which is the components provided in the arm they did not receive.

SUMMARY:
This study has two aims. The first is to understand more of what may be typical health trajectories after mass trauma for children and adults and what predicts these trajectories. The second is to understand what may be effective early interventions to prevent long-term health and psychosocial problems for youth (6-19). Participants are recruited from an outreach program implemented after a landslide killed 11 persons and destroyed 33 houses in Gjerdrum in Norway. One third of the inhabitants were evacuated. All evacuated are contacted and screened for trauma related difficulties. Those who have significant post-trauma reactions are offered trauma focused interventions.

DETAILED DESCRIPTION:
Two short step-wise interventions are developed for this study as an early intervention after mass trauma based on components from TF-CBT to test the relative importance of dosage and the sequencing of components.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to the landslide
* Between 6-19 years old
* A score of 15 or more on the CATS
* A score between 11 - 14 on the CATS and have additional problems that have started or worsened after the landslide.

Exclusion Criteria:

* Suicidal
* Psychotic

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
PTSD | Pre-treatment
  Measured with the Child and adolescent trauma screen (CATS). Range 0-60. Higher score means worse outcome.
PTSD | After 5 weeks
  Measured with the CATS (after 4-5 sessions)
PTSD | After 9 weeks
  Measured with the CATS (for those who continue to Step two)
PTSD | After 21 weeks
  Measured with the CATS
PTSD | After 33 weeks
  Measured with the CATS
PTSD | After 45 weeks
  Measured with the CATS
PTSD | After 57 weeks
  Measured with the CATS

SECONDARY OUTCOMES:
Depression | Pre-treatment
  Measured with Moods and feelings questionaire (MFQ-short). Range 0-13. Higher scores means worse outcome.
Depression | After 5 weeks
  Measured with MFQ-short
Depression | After 9 weeks
  Measured with MFQ-short
Depression | After 21 weeks
  Measured with MFQ-short
Depression | After 33 weeks
  Measured with MFQ-short
Depression | After 45 weeks
  Measured with MFQ-short
Depression | After 57 weeks
  Measured with MFQ-short

OTHER OUTCOMES:
Anxiety | Pre-treatment
  Measured with Screen for Child Anxiety Related Emotional Disorders (SCARED-5 Item)
Anxiety | After 5 weeks
  Measured with SCARED-5 Item
Anxiety | After 9 weeks
  Measured with SCARED-5 Item
Anxiety | After 21 weeks
  Measured with SCARED-5 Item
Anxiety | After 33 weeks
  Measured with SCARED-5 Item
Anxiety | After 45 weeks
  Measured with SCARED-5 Item
Anxiety | After 57 weeks
  Measured with SCARED-5 Item

CONTACTS AND LOCATIONS:
Overall Officials: Tine K Jensen, PhD, Principal Investigator — Norwegian Center for Violence and Traumatic Stress Studies
Locations (1):
- Norwegian center for violence and traumatic stress studies, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No